CLINICAL TRIAL: NCT03220711
Title: Study of Performance of Confocal Endomicroscope With Fluorescein Imaging Agent in the Colon
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study terminated due to equipment breakage and lack of funding.
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Danielle Kim Turgeon, Professor of Internal Medicine and Clinical Track Faculty Ombuds, Medical School, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: HUM00124968
Record Dates: First submitted 2017-07-14; First posted 2017-07-18 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Colonic Dysplasia; Adenomatous Polyps; Irritable Bowel Disease
MeSH Terms: conditions — Adenomatous Polyps; Irritable Bowel Syndrome | interventions — Fluorescein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subjects with abnormal colon tissue (Experimental): The study subjects will be high-risk for colonic adenomas (i.e. strong family history of adenomas/adenocarcinoma or personal history of adenomas/adenocarcinoma), known adenoma scheduled for endoscopic resection, or in subjects with suspected dysplasia in inflammatory bowel disease (IBD). Fluorescein will be sprayed on the area of interest to provide imaging contrast for the images taken with the confocal endomicroscope.
  Interventions: Device: confocal endomicroscope; Drug: Fluorescein

INTERVENTIONS:
Device: confocal endomicroscope — This instrument provides real-time endoscopic "histology" to guide endoscopic biopsy or endoscopic mucosal resection (EMR) in the patient study group during colonoscopies.
Drug: Fluorescein — Fluorescent dye used for imaging contrast only.
  Other Names: Fluorescite

SUMMARY:
The overall aim of this research project is to evaluate the imaging performance of a confocal endomicroscope. Fluorescein, an FDA-approved topical fluorescent dye, will be used to provide topical mucosal contrast. The purpose of this instrument is to provide real-time endoscopic "histology" to guide endoscopic biopsy or endoscopic mucosal resection (EMR) in the patient study group. This endomicroscope probe will be used during colonoscopies in subjects with colonic dysplasia, known colonic adenomatous polyps scheduled for endoscopic resection, or suspected dysplasia in subjects with Inflammatory Bowel Disease (IBD).

DETAILED DESCRIPTION:
The device is being tested in small groups of individuals: generally less than 10 for each of a variety of histologically different colonic lesions or diseases (eg. IBD, adenomas, sessile seriated adenomas (SSAs), hyperplastic polyps, normal tissue).

ELIGIBILITY:
Inclusion Criteria:

Subject meets at least one of the following criteria:

* At increased risk for colorectal cancer and colonic polyps
* Known colonic adenomas scheduled for colonic polyp resection
* Scheduled for outpatient colonoscopy for follow up surveillance of IBD with known dysplasia or who are at high risk for high grade dysplasia.

Exclusion Criteria:

Subject meets all of the following criteria:

* Subject is scheduled for outpatient colonoscopy in the Medical Procedures Unit at University of Michigan Health System.
* Subject is medically cleared for the procedure (e.g. washout for anticoagulants, co-morbidities) Standard practice guidelines for safely proceeding with the procedure will be sufficient for our study.
* Age 18 to 100 years
* Willing and able to sign informed consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2017-07-28 (Actual); Primary Completion 2022-06-02 (Actual); Study Completion 2022-06-02 (Actual)

PRIMARY OUTCOMES:
Depth-imaging capability of the confocal endomicroscope using an imaging contrast agent, fluorescein | five minutes
  The test product efficacy will be assessed by evaluating the fluorescence intensities measured from suspicious regions of colonic mucosa where the agent is administered compared to adjacent normal mucosa.

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Kim Turgeon, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States